CLINICAL TRIAL: NCT01790802
Title: A Multi-centre, Randomized Trial Into the Safety and Efficacy of Nanosecond Microsurgical Laser Intervention in Early Age-related Macular Degeneration
Brief Title: Laser Intervention in Early Age-Related Macular Degeneration Study
Acronym: LEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CERA201201; ACTRN12612000704897 (Registry Identifier: ANZCTR); CTN Number130/2012 (Other: TGA)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2018-07

CONDITIONS: Age-related Macular Degeneration
Keywords: laser treatment, high risk, early AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active laser (Experimental): Twelve 2RT nanosecond laser shots in two arcs of 6 shots superiorly and 6 shots inferiorly, inside the retinal vascular arcades at an approximate distance from the fovea of 3000 microns, with approximately one laser spot diameter between them.
  Interventions: Device: 2RT nanosecond laser
- Sham laser procedure (Sham Comparator): The maximum illumination button on hte 2RT laser will be briefly pressed by the operating physician at each of the 12 locations where and when the laser would normally be applied. The laser remains in standby mode preventing accidental laser firing.
  Interventions: Device: 2RT nanosecond laser

INTERVENTIONS:
Device: 2RT nanosecond laser — active laser therapy

SUMMARY:
The purpose of this study is to determine whether 2RT nanosecond laser therapy slows the progression to advanced age-related macular degeneration.

DETAILED DESCRIPTION:
LEAD is a patient and assessor masked, multi-centre randomized controlled exploratory medical device clinical investigation of 240 participants (1:1 active to shame laser procedure) designed to assess the effectiveness of nanosecond laser treatment of patients with early high-risk AMD.

No less than 240 participants will be randomized into either active laser treatment or sham laser procedure groups at a ratio of 1:1. Patient eligibility based on ocular inclusion criteria will be evaluated using measures of vision, fundus photography, OCT imaging, and macular integrity (MAIA) performed during the qualifying period. Fundus images and MAIA results will be sent to a coordinating centre where these will be reviewed to confirm eligibility based on lesion attributes and the criteria specified in the protocol. Following confirmation of eligibility by the coordinating centre, participants whom satisfy all the inclusion and exclusion criteria can be randomized. Allocation to treatment group will be stratified by smoking status. All participants will receive either active laser treatment or sham laser procedure at the treatment visit and be assessed for retreatment on a semi-annual basis. All participants will be contacted by telephone at 1 week and present for clinical examination visits at 1, 6, 12, 18, 24, 30 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 50 to 95 years of age at the time of consent
* Best corrected visual acuity (BCVA) of 6/12 (20/40) or better in each eye.
* Bilateral high-risk early AMD: At least one druse ≥125um within an inner macular zone (a circle with a radius of 1500 microns centred on the fovea) with or without pigment.
* A MAIA static threshold sensitivity less than 25 dB at any point, within a customized grid, as measured using a Macular Integrity Assessment (MAIA) device), at the same location of the one eye on two separate occasions.
* Pupil dilation of a least 5 mm in each eye
* Fundus photographs, optical coherence tomography (OCT) and fundus autofluorescence (FAF) images of adequate quality as assessed by the LEAD Image Reading Centre.
* Ability and willingness to consent, and be randomized, to the 2RT active or sham laser treatment, and all qualification and follow-up phases of the study.

Exclusion Criteria:

* Any evidence of definite geographic atrophy within the macula (a circle with a radius of 3000 microns centred on the fovea).
* Any black (hypofluorescent) area of FAF consistent with GA (roughly round or oval shape, sharp margins), and corroborated on colour photography as a patch of hypopigmentation.
* Any evidence of 'preclinical atrophy' as determined on OCT: loss of the outer retina (RPE and photoreceptors on the cube scan (Spectralis OCT) (49 horizontal B scans, 120 µm apart over a 20 x 20 degree scan). This covers approximately 6 x 6 mm in an emmetropic eye (N.B., peri-papillary atrophy (PPA) further than 1500 microns from the fovea is allowed).
* Current CNV, or past evidence of CNV in either eye.
* Any other experimental treatment for AMD, excluding dietary supplements, received in the past 12 months or thought likely to chronically change the course of the participant's retinal disease.
* Any OCT showing evidence of intraretinal fluid, or subretinal fluid for which CNV cannot be excluded as a cause.
* A subfoveal pigment epithelial detachment/drusenoid detachment greater than 1000 microns in diameter.
* Other macular disease with subretinal deposits not typical of AMD, e.g., Malattia Leventinese, Sorsby fundus dystrophy, Alports syndrome
* Ocular disease in either eye, other than AMD, which significantly compromises the ability to treat or visualize the fundus or would compromise the ability to assess any effect following laser application including;
* Known allergic hypersensitivity to fluorescein.
* Previous retinal or other ocular surgical procedures, the effects of which may now or in the future complicate assessment of the progression of AMD.
* Requirement for any systemic or ocular medication known to be toxic to the retina, such as: Deferoxamine, Chloroquine/Hydroxychloroquine (Plaquenil), Chlorpromazine, Phenothiazines, Ethambutol
* Any serious systemic disease that will preclude a 3 year survival and regular attendance for follow up.
* Sensitivity to contact lens application.
* Any condition that would make adherence to the examination schedule for 3 years difficult or unlikely.
* Any history of prior laser surgery to the retina.
* Intraocular pressures of 26mm Hg or higher or if there is some reason to believe the participant may have glaucoma
* Significant cataract: Nuclear cataract grade 2 or 3, cortical cataract Grade 2 or 3 or posterior subcapsular cataract Grade 2 or 3, by Simplified Cataract Grading System (WHO Cataract Grading Group).

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
progression to advanced Age-related Macular Degeneration (AMD) in the treated eye | 36 months
  rate of progression to advanced AMD, either Choroidal Neovascularization (CNV), Geographic Atrophy (GA) or preclinical atrophy, in the study eye of treatment group compared to the sham procedure group

SECONDARY OUTCOMES:
progression to advanced AMD in the untreated eye | 36 months
  rate of progression to advanced AMD, CNV, GA or preclinical atrophy in the fellow (untreated) eye

OTHER OUTCOMES:
reversal of early clinical indicators of AMD | 36 months
  reversal of early clinical indicators of AMD (drusen area)
Improvements in visual acuity | 36 months
  improvement in VA

CONTACTS AND LOCATIONS:
Overall Officials: Robyn H Guymer, PhD, FRANZCO, Study Chair — Deputy Director CERA
Locations (1):
- Centre for Eye Research Australia - Royal Victorian Eye & Ear Hospital, East Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Goh KL, Wintergerst MWM, Abbott CJ, Hadoux X, Jannaud M, Kumar H, Hodgson LAB, Guzman G, Janzen S, van Wijngaarden P, Finger RP, Guymer RH, Wu Z. HYPERREFLECTIVE FOCI NOT SEEN AS HYPERPIGMENTARY ABNORMALITIES ON COLOR FUNDUS PHOTOGRAPHS IN AGE-RELATED MACULAR DEGENERATION. Retina. 2024 Feb 1;44(2):214-221. doi: 10.1097/IAE.0000000000003958. PMID 37831941
- [Derived] Wu Z, Luu CD, Hodgson LAB, Caruso E, Chen FK, Chakravarthy U, Arnold JJ, Heriot WJ, Runciman J, Guymer RH; LEAD Study Group. USING MICROPERIMETRY AND LOW-LUMINANCE VISUAL ACUITY TO DETECT THE ONSET OF LATE AGE-RELATED MACULAR DEGENERATION: A LEAD Study Report. Retina. 2021 May 1;41(5):1094-1101. doi: 10.1097/IAE.0000000000002982. PMID 33009222